CLINICAL TRIAL: NCT04786847
Title: A Phase 1 Safety, Tolerability, Biodistribution, Dosimetry and Efficacy Study of 177Lu-DOTA-TLX591 With Best Standard of Care in Patients With PSMA Expressing Metastatic Castration-resistant Prostate Cancer
Brief Title: 177Lu-DOTA-TLX591 Safety, Biodistribution and Dosimetry Study
Acronym: ProstACTSelect
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Telix Pharmaceuticals (Innovations) Pty Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 177Lu-TLX591-001
Record Dates: First submitted 2021-02-24; First posted 2021-03-08 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Metastatic Prostate Cancer
Keywords: prostate cancer; biodistribution; 177Lu-DOTA-TLX591; pharmacokinetics; dosimetery; safety; preliminary efficacy; standard of care; gallium-68 labeled PSMA-11 (68Ga-PSMA-11) PET/CT scan; novel androgen axis drug
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Approximately 50 eligible patients will be enrolled and evaluated for safety and tolerability as well as undergo imaging to allow determination of the biodistribution and dosimetry 177Lu-DOTA-TLX591. Twenty-five patients will also be enrolled in a biodistribution and dosimetry sub-study, involving the collection of quantitative single-photon emission computerized tomography (SPECT) or single-photon emission computerized tomography/computerized tomography (SPECT/CT) data in a subset of patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single administration of 177Lu-DOTA-TLX591 (Experimental): Two single IV infusions of 76 mCi (2.8 GBq) each (equivalent to a 45 mCi/m2 administered activity in a standard 1.7m2 individual) of 177Lu-DOTA-TLX591, given 14 days apart. This therapy will be administered with the current standard of care treatment regimens.
  Interventions: Biological: 177Lu-DOTA-TLX591

INTERVENTIONS:
Biological: 177Lu-DOTA-TLX591 — TLX591, a monoclonal antibody HuX591 conjugated with a DOTA chelator and radiolabelled with 177Lu (177Lu-TLX591)

SUMMARY:
This is a Phase 1 trial of TLX591, a monoclonal antibody HuX591 conjugated with a DOTA chelator and radiolabelled with 177Lu (177Lu-DOTA-TLX591). TLX591 is being developed as a PSMA-targeting antibody to be radiolabelled with a therapeutic radiosotope for the treatment of PSMA-expressing tumours, therefore this study has been designed to assess the safety and tolerability, pharmacokinetics, whole body biodistribution and radiation dosimetry of 177Lu-DOTA-TLX591.

DETAILED DESCRIPTION:
This multi-center prospective Phase 1 study is designed to evaluate the safety, tolerability, biodistribution and dosimetry of 177Lu-DOTA-TLX591 administered to patients together with best SoC with metastatic castration-resistant prostate cancer (mCRPC) that expresses PSMA and has progressed despite prior treatment with a novel androgen axis drug (NAAD).

PSMA positivity will be defined by 68Ga-PSMA-11 or [18F]DCFPyL PET/CT where at least one site of metastatic disease has an intensity of tracer uptake significantly greater than normal liver (i.e., standardized uptake value [SUV]max at least 1.5 times SUV of normal liver.

Approximately 25-50 eligible patients will be enrolled and evaluated for safety and tolerability as well as undergo imaging to allow determination of the biodistribution and dosimetry 177Lu-DOTA-TLX591. All patients will receive two single intravenous (IV) infusions of 76 mCi each (equivalent to 45 mCi/m2 in a standard 1.7m2 individual) of 177Lu-DOTA-TLX591, given notionally 14 days apart, plus best SoC.

Twenty-five patients will also be enrolled in a biodistribution and dosimetry sub-study, involving the collection of quantitative single-photon emission computerized tomography (SPECT) or single-photon emission computerized tomography/computerized tomography (SPECT/CT) data in a subset of patients.

SPECT/CT scans will be performed after administration of the drug, at the following timepoints: i) 4h ± 5 min, ii) 24 ± 4h, iii) 96 ± 4h, iv) Day 7± 4h and v) Day 13± 4h. These SPECT/CT scans will be conducted to further support safety monitoring and to understand exposure of tumour and healthy tissue to 177Lu-DOTA-TLX591.

Imaging data from the first five patients enrolled in the biodistribution study will be analysed and, if appropriate, the number of imaging timepoints will be reduced to three for subsequent patients. Qualitative comparison of 68Ga-PSMA-PET/CT images and 177Lu-DOTA-TLX591 images will also be undertaken for patients undergoing the biodistribution study to ensure equivalence of radiopharmaceutical localization to tumour sites and equivalent off-target localization.

Blood samples for pharmacokinetic analysis will be performed at 15 min ± 5 min before administration of the drug, and at the following timepoints after dosing: i) end of infusion ± 5min, ii) 60 min ± 5 min, ii) 4h ± 5 min, iii) 24 ± 4h, v) 48 ± 4h, vi) 96 ± 4h, vii) Day 7± 4h and viii) Day 13± 4h.

Collection of information on prior and concomitant medications and adverse events (AEs), as well as the review of temporary contra-indications and conditions for withdrawal, will occur at every patient interaction.

ELIGIBILITY:
Inclusion Criteria:

* Be male, at least 18 years old, with histologically/pathologically confirmed metastatic adenocarcinoma.
* Be of ECOG Performance Status 0, 1, or 2 and have an estimated life expectancy of ≥ 6 months.
* Have metastatic disease (≥1 metastatic lesions present on baseline whole body CT, MRI, or bone scintigraphy).
* Have castration-resistant PC (defined as disease progressing despite castration by orchiectomy or ongoing use of luteinizing hormone-releasing hormone [LHRH] agonists) and must have a castrate level of serum/plasma testosterone (< 50 ng/dL or <1.7 nmol/L).
* In the mCRPC setting, must have received a minimum of 12 weeks of prior therapy with a NAAD, either enzalutamide or abiraterone plus prednisone.
* Have received one line of prior taxane therapy, or have refused or are ineligible for taxanes
* Have disease that is progressing at study entry, despite a castrate testosterone level (<50 ng/dL or <1.7 nmol/L), by the demonstration of at least one of the following:

  1. Increase in PSA greater than 25% and > 2 ng/mL above nadir, confirmed by progression at 2 timepoints at least 3 weeks apart.
  2. Progressive disease or new lesion(s) (relative to previous imaging) in the viscera or lymph nodes as per RECIST1.1 or in bone as per Prostate Cancer Working Group 3 [PCWG3). Any ambiguous results are to be confirmed by additional imaging modality (e.g., CT, Tc-99m bone scintigraphy)
* Have disease which is PSMA positive, as demonstrated by a 68Ga-PSMA-11 PET/CT or [18F]DCFPyL PET/CT scan and confirmed as eligible by local reader (patient must have at least one site of metastatic disease with SUVmax ≥1.5 times the SUV of normal liver). If the disease meets the criteria for PSMA positivity, but there is one or more soft tissue lesion of ≥2 cm that is not PSMA positive, then the patient is to be excluded on the grounds that there is substantial disease which might not respond to the therapy.
* Must have recovered to ≤ Grade 2 from all clinically significant toxicities related to prior therapies (i.e., surgery, local radiotherapy, NAAD, chemotherapy, etc.).
* Can be receiving a bisphosphonate or denosumab regimen provided tolerance to this therapy has been proven.

  11. Have adequate organ function at Screening:

  a. Bone marrow: i. Platelets ≥150×109/L ii. Absolute neutrophil count >1.5×109/L iii. Hemoglobin ≥10g/dL (no red blood cell transfusion in the previous 4 weeks) b. Liver function: i. Total bilirubin ≤1.5×the upper limit of normal (ULN). For patients with known Gilbert's Syndrome ≤3×ULN is permitted ii. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≤3×ULN OR ≤5×ULN for patients with liver metastases c. Renal function: i. Serum/plasma creatinine ≤1.5×ULN or creatinine clearance ≥50 mL/min
* Have the capacity to understand the study and be able and willing to comply with all protocol requirements.
* Must comply with the radiation protection guidelines (including hospital admissions and isolation) that are applied by the treating institution in order to protect their contacts and the general public.
* Must agree to practice adequate precautions to prevent pregnancy in a partner and to avoid potential problems associated with radiation exposure to the unborn child (Refer to Clinical Trials Facilitation Group, 2020: Recommendations related to contraception and pregnancy testing in clinical trials Version 1.1, CTFG, 2020).

Exclusion:

* Are unable, in the opinion of the Investigator, to understand or are unwilling to sign a written informed consent document or to follow investigational procedures.
* Have PC with pathological findings consistent with small cell or any histology other than adenocarcinoma of the prostate. If there are minor elements of neuroendocrine histology, this is acceptable.
* Experiencing uncontrolled pain
* Diagnosed with other malignancies that are expected to alter life expectancy or may interfere with disease assessment. Patients with a prior history of malignancy that has been adequately treated and who have been disease-free for more than 3 years are eligible, as are patients with adequately treated non-melanoma skin cancer, and superficial bladder cancer.
* At increased risk of hemorrhage, or with a recent history of a thrombotic event (e.g., deep vein thrombosis [DVT]/ pulmonary embolism [PE]) and/or are using long-term anti-coagulant or anti-platelet agents.
* Have received prior administration of monoclonal antibody (mAb) J591 or HuJ591 or any other PSMA targeted therapy.
* Have known allergies, hypersensitivity, or intolerance to the investigational drug or its excipients.
* Have received systemic anti-cancer therapy (e.g., chemotherapy, immunotherapy, or biological therapy) and/or radiation therapy within 4 weeks of enrollment OR if any significant AEs have not resolved to National Cancer Institute (NCI) AE Criteria ≤2; OR are receiving other concurrent cytotoxic chemotherapy, immunotherapy, radioligand therapy, or investigational therapy.
* Have received prior treatment with radiopharmaceuticals containing, but not limited to, the following radioisotopes: 89Strontium, 153Samarium, 186Rhenium, 188Rhenium, 223Radium; or have received hemi-body irradiation within 6 months prior to randomization.
* Have received other investigational agents within 4 weeks of randomization.
* Have known brain metastases (any size) or hepatic metastases > 1 cm.
* Have a history of seizure and/or stroke within past 6 months.
* Have clinical or radiologic findings indicative of impending cord compression or experiencing symptomatic cord compression.
* Have a serious active or sub-clinical infection, or angina pectoris or heart failure (New York Heart Association [NYHA] Class III or IV), significantly prolonged QT interval or other serious illness(es) involving the cardiac, respiratory, central nervous, renal, hepatic or hematological organ systems, which might impair the ability to complete this study or could interfere with determination of causality of any adverse effects experienced in this study, or which require treatment that could interact with study treatment.
* Have received treatment with any PARP inhibitors (i.e., Olaparib) or with any platinum based anti-neoplastic drugs.
* Have a known alteration in breast cancer genes (BRCA) BRCA1, BRCA2, or Ataxia Telangiectasia Mutated Gene (ATM) gene and are eligible to receive Olaparib therapy according to their treating institution SoC.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-01-30 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v5.0 | Day 1 to 5 years
  To monitor the safety and tolerability of molecularly targeted radiotherapy with 177Lu-DOTA-TLX591, administered in two cycles in combination with best SoC in patients with PSMA-expressing metastatic castrate resistant prostate cancer.
  Treatment emergent adverse events (TEAE) will be classified according to MedDRA (Medical Dictionary for Regulatory Activities), frequency, severity according to NCI CTCAE V5.0, seriousness, and relationship of study treatment will be assessed. Laboratory abnormalities will be assessed according to the NCI CTCAE v.5.0.

SECONDARY OUTCOMES:
Whole body and organ uptake of 177Lu-DOTA-TLX591 | Day 1 to Day 15
  Quantitate the absorbed radiation doses (expressed as Gy/MBq) of administered 177Lu-DOTA-TLX591) to kidneys, liver, lungs, spleen, bone/red marrow and salivary glands below acceptable safe limits as defined by ARPANSA
Compare the whole body and organ uptake of 177Lu-TLX591 and 68Ga-PSMA-11 radioactive tracers | Day 1 to 15
  Qualitatively equivalent biodistribution of 68Ga-PSMA-11 and 177Lu-DOTA-TLX591, as determined by image interpretation by expert radiologist or nuclear medicine physician.

CONTACTS AND LOCATIONS:
Locations (3):
- Australia (3):
  - GenesisCare Newcastle, Newcastle, Gateshead
  - Diagnostic Nuclear Imaging at Hollywood Private Hospital, Perth, Western Australia
  - GenesisCare SJOg Medical Centre,Murdoch, Perth, Western Australia

IPD SHARING:
Plan to Share IPD: No